CLINICAL TRIAL: NCT06266832
Title: The Efficacy and Safety of Short-course Radiation Combined With Adebrelimab and CAPEOX Neo-adjuvant Therapy for Organ-retention in Patients With MSS/pMMR Ultra Low Rectal Adenocarcinoma: A Prospective, Single-arm Study
Brief Title: The Efficacy and Safety of Short-course Radiation Combined With Adebrelimab and CAPEOX Neo-adjuvant Therapy for Organ-retention in Patients With MSS/pMMR Ultra Low Rectal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230727
Record Dates: First submitted 2024-01-28; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total Neoadjuvant Therapy with Short-course Radiation followed by Adebrelimab plus CAPEOX (Experimental): The enrolled patients with MSS-type advanced ultra low rectal adenocarcinoma will receive a combined regimen of neoadjuvant chemoradiotherapy combined with immunotherapy and biopsy or local excision.
  Radiotherapy uses a short-range mode, irradiating the primary tumor and high-risk areas with dose of 25 Gy.
  After radiotherapy, PD-L1 antibody (20mg/kg, intravenously guttae, 2courses) immunotherapy combined with 2 courses of CAPEOX chemotherapy was performed.
  1-4 weeks after the end of the combined treatment plan in step 2), biopsy or local excision of the lesion is performed.
  Interventions: Drug: Adebrelimab; Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Short-course Radiation; Procedure: Biopsy

INTERVENTIONS:
Drug: Adebrelimab — This product is administered by intravenously guttae. The recommended dose of subcutaneous injection is 20mg/kg, administered every 3 Weeks (Q3W).
  Other Names: SHR-1316
Drug: Oxaliplatin — 130mg/m2, ivgtt, d1, Q3W
Drug: Capecitabine — 1000mg/m2, po, bid, d1-14, Q3W
Radiation: Short-course Radiation — Short-course radiotherapy, using three-dimensional conformal or intensity-modulated radiotherapy, the dose is divided into 5Gy/f, the total dose is 25Gy/5f, 1f/d, and the irradiation is completed within 7 days.
Procedure: Biopsy — local excision or TME surgery (total mesorectal excision) Biopsy can choose endoscopic or needle biopsy, colcal excision refers to excison of the local lession after total neoadjuvant therapy. The total mesorectal excision can choose open, laparoscopic or robotic according to the specific condition of the patient.

SUMMARY:
To evaluate the efficacy, safety and organ retention rate of short-course radiation combined with Adebrelimab and CAPEOX neoadjuvant therapy in patients with MSS/pMMR ultra low rectal adenocarcinoma.

DETAILED DESCRIPTION:
At present, neoadjuvant chemoradiotherapy (nCRT) combined with total mesorectal excision (TME) is the main standard treatment, and the choice of treatment modalities is limited. The emergence of immunotherapy has provided a new direction for the exploration of neoadjuvant therapy for rectal adenocarcinoma. At the same time, a number of studies have also shown that appropriate radiotherapy intensity can promote immune response. Therefore, the investigators intend to conduct the clinical trail to explore the effect of short-course radiotherapy combined with PD-L1 combined and chemotherapy as TNT (total neoadjuvant therapy) on organ retention rate in patients with With MSS/pMMR Ultra Low Rectal Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to receive neoadjuvant therapy.
2. ≧18 years old.
3. Diagnosed by digital rectal examination, colonoscopy, and high-resolution MRI of the pelvis, the tumor is less than or equal to 5 cm from the anus.
4. Histologically diagnosed as rectal adenocarcinoma.
5. MMR protein detection or MSI gene detection of rectal cancer specimens confirmed pMMR or MSS before treatment .
6. The clinical staging by pelvic contrast-enhanced CT and pelvic high-resolution MRI were stage I, II and III.
7. The patient has good compliance and can come to the hospital for re-examination as required.
8. ECOG Scale of Performance Status score 0-1 point.
9. Have not received anti-tumor and immunotherapy before enrollment.
10. Laboratory inspections must meet the following standards:

    1. White blood cell count>3.5×109/L, absolute value of neutrophils>1.8×109/L, platelet count ≥75×109/L, hemoglobin ≥100g/L;
    2. INR≤1.5, and APTT≤1.5 times the upper limit of normal or partial prothrombin time (PT) ≤1.5 times the upper limit of normal;
    3. Total bilirubin ≤ 1.25 times the upper limit of normal; ALT and AST < 5 times the upper limit of normal;
    4. 24h creatinine clearance >50mL/min or serum creatinine <1.5 times the upper limit of normal.
11. Voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

1. History of other malignant diseases other than rectal cancer in the past 5 years.
2. Patients with metastases from other sites (stage IV patients).
3. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. requiring emergency surgery.
4. Known allergic to oxaliplatin, capecitabine, Adebrelimab and other drugs.
5. Pathologically suggested signet ring cell carcinoma and mucinous adenocarcinoma.
6. dMMR or MSI-H patients.
7. The patient is accompanied by any unstable systemic disease, including but not limited to: severe infection, uncontrolled diabetes, hypertension uncontrolled by medication, unstable angina, cerebrovascular accident or transient cerebral ischemia, myocardial Infarction, congestive heart failure, severe cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease; disease affecting the patient's life.
8. The disease (such as mental illness, etc.) or condition (such as alcoholism or drug abuse, etc.) associated with the patient will increase the risk of the patient receiving the trial drug treatment or affect the patient's compliance with the trial requirements, or may confuse the research results.
9. Active autoimmune disease that may worsen while receiving immunostimulants.
10. Known history of positive HIV test or known acquired immunodeficiency syndrome.
11. Patients who are using immunosuppressive agents, except for the following conditions:

    1. Intranasal, inhaled, topical steroids, or topical steroid injections (eg, intra-articular injections);
    2. Physiological doses of systemic corticosteroids ≤10 mg/day prednisone or equivalent; 3) Steroids used to prevent allergic reactions (eg, before CT scan).
12. Received any other experimental drug treatment or participated in another interventional clinical trial within 30 days before screening.
13. Women who are pregnant or breastfeeding or who plan to become pregnant or breastfeeding during the study period; men or women who are unwilling to take effective contraceptive measures.
14. Vulnerable groups, including mentally ill, cognitively impaired, critically ill patients, minors, etc.
15. Other conditions that the investigator judges that the patient is not suitable to participate in the clinical study, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Organ retention rate | After 2 weeks (once biopsy or local excision is done)
  population who achieve complete clinical response after total neoadjuvant therapy

SECONDARY OUTCOMES:
Total mesorectal excision rate | After 2 weeks (once biopsy or local excision is done)
  population who not achieve complete clinical response after total neoadjuvant therapy
Total mesorectal excision rate after recurrence | from primary evaluation at 2 weeks after total neoadjuvant therapy finished
  population who recurrent and have Salvage total mesorectal excision after achieving complete clinical response after total neoadjuvant therapy
Tumor regression grade | After 2 weeks (once biopsy or local excision is done)
  Tumor regression grade following short-course radiation then Envafolimab Plus CAPEOX as assessed by AJCC/CAP TRG system
Overall survival | Up to 3 years
  The proportion of participants who remain survival at 3 years
Disease free survival | Up to 3 years
  The time from randomization to the first event of either recurrent disease or death
TRAEs | Up to 3 years
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0
QoL | Up to 3 years
  Quality of life of the patients in total neoadjuvant settings of short-course radiation followed with Adebrelimab Plus CAPEOX as assessed by Functional Assessment of Cancer Therapy - Colorectal (FACT-C) questionnaire liscenced from The Functional Assessment of Chronic Illness Therapy System ("FACIT System"). By using the Manual scoring template, some items are reverse scored. Subscale scores, total scores and TOI scores. The higher the score, the better the QOL.

CONTACTS AND LOCATIONS:
Overall Officials: sheng dai, MD&PhD, Principal Investigator — China, Zhejiang Sir Run Run Shaw Hospital, Zhejiang University School of Medicine
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No